CLINICAL TRIAL: NCT05437315
Title: GD2/PSMA Bi-specific CAR-T Cells For the Treatment of GD2 and PSMA Positive Solid Tumors
Brief Title: GD2/PSMA Bi-specific CAR-T Cell Therapy
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shenzhen Geno-Immune Medical Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GIMI-IRB-22003
Record Dates: First submitted 2022-06-21; First posted 2022-06-29 (Actual); Last update posted 2022-06-29 (Actual); Status verified 2022-06

CONDITIONS: Solid Tumor
Keywords: CAR-T; Solid tumor; GD2; PSMA

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- bi-4SCAR-GD2/PSMA T Cell Therapy for GD2 and PSMA positive tumor (Experimental)
  Interventions: Biological: bi-4SCAR GD2/PSMA T cells

INTERVENTIONS:
Biological: bi-4SCAR GD2/PSMA T cells — Infusion of bi-4SCAR GD2/PSMA T cells at 10^6 cells/kg body weight via IV

SUMMARY:
The purpose of this clinical trial is to assess the feasibility, safety and efficacy of anti-GD2/PSMA bi-specific CAR-T cell therapy in patients with GD2 and PSMA positive tumor. Another goal of the study is to learn more about the function of the anti-GD2/PSMA bi-specific CAR-T cells and their persistency in patients.

DETAILED DESCRIPTION:
Patients with refractory and/or recurrent solid tumors have poor prognosis despite complex multimodal therapy; therefore, novel curative approaches are needed. The investigators are attempting to use T cells obtained directly from the patient, which can be genetically modified to express a 4th generation anti-GD2/PSMA bi-specific chimeric antigen receptor (bi-4SCAR-GD2/PSMA). The chimeric antigen receptor (CAR) molecules enable the T cells to recognize and kill tumor cells through the recognition of a surface antigen, GD2 or PSMA, which is expressed at high levels on tumor cells but not at significant levels on normal tissues.

Disialoganglioside (GD2) is a well-studied tumor associated antigen which is expressed uniformly in nervous system-related tumors but at low levels in normal tissues. Over the past few years, CAR-T therapy against GD2 in tumor has achieved encouraging but modest outcomes. Only a fraction of patients achieved measurable responses. In solid tumors, GD2 CAR-T therapy alone may not as effective as CAR-T cell therapy in hematological malignancies.

Prostate-specific membrane antigen (PSMA) is expressed in normal prostate and upregulated in prostate tumor. Therefore, PSMA is a promising target for immunotherapy of prostate cancer. However, PSMA is not restricted to prostate cancer and it is known that PSMA is enriched in the tumor stromal environment. Based on immunostaining, it is confirmed that PSMA is expressed in a variety of solid tumors, including brain tumor, neuroblastoma and some lymphomas.

To overcome tumor escape of single target antigen and enhance in vivo CAR-T efficacy, a novel bi-specific GD2/PSMA CAR-T therapy regimen is developed to include booster and consolidation CAR-T applications to target highly-refractory cancer. The aim is to evaluate safety and long term efficacy of the bi-CAR-T therapy strategy in GD2 and/or PSMA positive cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with tumors have received standard first-line therapy and have been judged to be non-resectable, metastatic, progressive or recurrent.
2. The expression status of GD2 or PSMA antigens in the tumor tissue will be determined for eligibility. Positive expression is defined by GD2 and PMSA antibody staining results based on immunohistochemistry or flow cytometry analyses.
3. Body weight greater than or equal to 10 kg.
4. Age: ≥1 year and ≤ 75 years of age at the time of enrollment.
5. Life expectancy: at least 8 weeks.
6. Prior Therapy:

   There is no limit to the number of prior treatment regimens. Any grade 3 or 4 non-hematologic toxicity of any previous therapy must be resolved to grade 2 or less.
7. Participant must not have received hematopoietic growth factors for at least 1 week prior to mononuclear cells collection.
8. At least 7 days must have elapsed since the completion of therapy with a biologic agent, selected targeted agent or a metronomic non-myelosuppressive regimen.
9. At least 4 weeks must have elapsed since prior therapy that included a monoclonal antibody.
10. At least 1 week since any radiation therapy at the time of study entry.
11. Karnofsky/jansky score of 60% or greater.
12. Cardiac function: Left ventricular ejection fraction greater than or equal to 40/55 percent.
13. Pulse Ox greater than or equal to 90% on room air.
14. Liver function: defined as alanine transaminase (ALT) <3x upper limit of normal (ULN), aspartate aminotransferase (AST) <3x ULN; serum bilirubin and alkaline phosphatase <2x ULN.
15. Renal function: Patients must have serum creatinine less than 3 times upper limit of normal.
16. Marrow function: White blood cell count ≥1000/ul, Absolute neutrophil count ≥500/ul, Absolute lymphocyte count ≥500/ul, Platelet count ≥25,000/ul (not achieved by transfusion).
17. Patients with known bone marrow metastatic disease will be eligible for study as long as they meet hematologic function criteria, and the marrow disease does not have hematologic toxicity.
18. For all patients enrolled in this study, themselves or their parents or legal guardians must sign an informed consent and assent.

Exclusion Criteria:

1. Existing severe illness (e.g. significant cardiac, pulmonary, hepatic diseases, etc.) or major organ dysfunction, or greater than grade 2 hematologic toxicity.
2. Untreatable central nervous system (CNS) metastasis: Patients with previous CNS tumor involvement that has been treated and is stable for at least 6 weeks following completion of therapy are eligible.
3. Previous treatment with other genetically engineered GD2 or PSMA-specific CAR T cells or antibody therapy.
4. Active HIV, Hepatitis B virus (HBV), Hepatitis C virus (HCV) infection or uncontrolled infection.
5. Patients who require systemic corticosteroid or other immunosuppressive therapy.
6. Evidence of tumor potentially causing airway obstruction.
7. Inability to comply with protocol requirements.
8. Insufficient CAR T cells availability.

Ages: 1 Year to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-06-30 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of patients with adverse events. | 6 months
  Determine the toxicity profile the bi-4SCAR GD2/PSMA cells with Common Toxicity Criteria for Adverse Effects version 4.0

SECONDARY OUTCOMES:
Anti-tumor effects | 1 year
  Objective complete response (CR) are assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria.
Anti-tumor effects | 1 year
  Objective partial response (PR)) are assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria.
The persistence of bi-4SCAR GD2/PSMA T cells | 1 year
  Scale of tumor burden
The expansion bi-4SCAR GD2/PSMA T cells | 1 year
  Scale of CAR copies
Survival time of the patients | 3 years
  The progression free survival (PFS) time of the patients treated with the bi-4SCAR GD2/PSMA T cells will be evaluated
Survival time of the patients | 3 years
  The overall survival (OS) time of the patients treated with the bi-4SCAR GD2/PSMA T cells will be evaluated

CONTACTS AND LOCATIONS:
Locations (1):
- Shenzhen Geno-immune Medical Institute, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No